CLINICAL TRIAL: NCT00299416
Title: Combined Neuroprotective Modalities Coupled With Thrombolysis in Acute Ischemic Stroke: A Pilot Study of Caffeinol and Mild Hypothermia
Brief Title: Caffeinol Hypothermia Protocol
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Responsible Party: James C. Grotta, MD-, UT- Houston Health Science Center, Department of Neurology
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HSC- MS-02-188; P50NS44277 project #1
Record Dates: First submitted 2006-03-02; First posted 2006-03-06 (Estimated); Results first posted 2011-05-03 (Estimated); Last update posted 2011-05-03 (Estimated); Status verified 2011-04

CONDITIONS: Acute Ischemic Stroke
Keywords: Stroke; Nonhemorrhagic; hypothermia
MeSH Terms: conditions — Ischemic Stroke; Stroke; Hypothermia | interventions — caffeinol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Caffeinol — Infusion of caffeinol (9mg/kg caffeine + 0.4g/kg ethanol) over 2 hours.
Procedure: hypothermia — External or internal cooling for 24 hours and rewarming over 12 hours.

SUMMARY:
Caffeinol is a combination of caffeine and alcohol. The amount given is about the same as 1-2 glasses of wine and 3-4 cups of coffee. The patient receives a one time dose given over two hour while being cooled to 34.5 C.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-80 years
2. Clinical presentation of acute ischemic stroke
3. Computed tomography (CT) scan compatible with acute ischemic stroke.
4. Time to caffeinol treatment < 240 minutes from stroke onset.
5. Time to hypothermia initiation < 300 minutes from stroke onset.
6. Presumed cortical location of stroke (must have at least on sign such as aphasia, neglect, visual field cut)
7. National Institutes of Health Stroke Scale (NIHSS) > 8 at time of each treatment.
8. Tissue plasminogen activator (TPA) treated patients must meet all established criteria for TPA.

Exclusion Criteria:

1. Etiology other than ischemic stroke.
2. Item 1a on NIHSS > 1
3. Signs/symptoms of subcortical, brainstem or cerebellar stroke.
4. Symptoms resolving or NIHSS < 8 at time of each treatment.
5. NIHSS > 20 if right hemisphere or >25 if left hemisphere
6. Known alcoholic
7. Clinical or laboratory evidence of alcohol intoxication.
8. Historical evidence of exogenous caffeine exposure beyond daily consumption of coffee or soft drinks.
9. Known hematologic dyscrasias that affect thrombosis.
10. Comorbid conditions likely to complicate therapy:

    1. End-stage cardiomyopathy
    2. Uncompensated or clinically significant arrhythmia
    3. Myopathy
    4. Liver disease
    5. History of pelvic or abdominal mass likely to compress inferior vena cava.
    6. End-stage AIDS
    7. History of clinically significant gastrointestinal (GI) bleeding
    8. Impaired renal function with creatinine clearance, 50 ml/min
11. Intracerebral / intraventricular hemorrhage
12. Systolic blood pressure (SBP) > 210 or < 100; diastolic blood pressure (DBP) > 100 or < 50 mmHg
13. Severe coagulopathy
14. Pregnancy
15. Use of monoamine oxidase inhibitor (MAOI),serotonin-specific reuptake inhibitor (SSRI) or Tricyclic Antidepressants (TCA) within the preceding 2 weeks
16. Known history of epilepsy.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2003-02; Primary Completion 2009-01 (Actual); Study Completion 2009-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James C. Grotta, MD, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- Memorial Hermann Hospital - Medical Center, Houston, Texas, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patient/& or family was approached by one of the investigators in the Emergency Department in order to obtain informed consent.
Pre-assignment Details: Open label pilot trial; Caffeinol Arm
Groups:
- Caffeinol: Caffeinol will be administered over a 2 hour infusion period. Dosage of caffeinol is based on on-going dose escalation trials and based on the patients weight. Currently the dosage is: ethanol 10% (0.4gm/kg) and caffeine 9 mg/kg.
Period: Overall Study
Arm/Group | Caffeinol
Started | 30
Completed | 30
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Caffeinol
Number analyzed (Participants) | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 28
  >=65 years | 2
Age Continuous [Mean (Standard Deviation); unit: years] | 54.7 (15.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18
  Male | 12
Region of Enrollment [Number; unit: participants]
  United States | 30

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Symptomatic Intracerebral Hemorrhage
Description: Symptomatic intracerebral hemorrhages were measured by a full NIHSS(National Institute of Health Stroke Scale) prior to caffeinol & hypothermia,at the end of hypothermia & rewarming, 24 hrs after stroke onset, daily during hospitalization,& at the 90 day follow-up visit. In addition, modified NIHSS were done hourly during the 24 hr hypothermia period & 12 hr rewarming period. At the end of rewarming an MRI was obtained to verify if hemorrhages or neurologic deteriorations were present.NIHSS scores severity of stroke on 11 items;more points given for greater deficiencies(range 0-42,0=normal)
Time Frame: from pre-dosage to 90 day followup
Population: Number of participants were determined by intention to treat. We did not use any imputation technique.
Measure: Number; unit: participants
Arm/Group | Caffeinol
Number analyzed (Participants) | 30
participants | 0

2. Secondary Outcome: Feasibility: Time Required to Reach the Target Core Temperature or Lowest Tolerated Temperature, Stability of Patient Temperature, Control of Rewarming,
Description: Hypothermia will be maintained for 24 hours, afterward, the patient will be rewarmed, gradually, over 12 hours to 36.5C.
Time Frame: rewarming over 12 hours until 36.5C has been achieved
Reporting Status: Not Posted
Measure: Number; unit: participants with acute ischemic stroke

3. Secondary Outcome: Achievement of Therapeutic Serum Ethanol and Caffeine Levels, and Amount of Sedation Needed to Suppress Shivering.
Time Frame: rewarming over 12 hours until 36.5C has been achieved
Reporting Status: Not Posted
Measure: Number; unit: participants with acute ischemic stroke

4. Secondary Outcome: Efficacy: NIHSS < 2 at 24 Hours, Modified Rankin Scale (mRS) < 2 at 3 Months, NIHSS < 2 at 3 Months, and Length of Hospital and ICU Stay.
Description: NIHSS score of ≤ 2 24 hours after stroke onset modified Rankin Scale (mRS) < 2 at 90 day followup NIHSS score of ≤ 2 at daily duration of hospitalization and ICU stay and 90 day follow up.
Time Frame: 90 days
Reporting Status: Not Posted
Measure: Number; unit: participants with acute ischemic stroke

5. Primary Outcome: Number of Participants With Catheter Related Complications During Hypothermia & Rewarming
Description: Catheter-related complications assessed whether participants had bleeding (major hemorrhaging) that required a blood transfusion, this was determined by labs. Participants were monitored for infections every hour during vital signs in the 24 hour hypothermia phase and 12 hour rewarming phase.
Time Frame: over 36 hour period
Measure: Number; unit: participants
Arm/Group | Caffeinol
Number analyzed (Participants) | 30
participants | 0

6. Primary Outcome: Number of Participants With Cardiorespiratory Failure
Description: The possibility of cardiorespiratory failure was monitored every 30 minutes during the 24 hour hypothermia period based on vitals signs and oxygen saturation.
Time Frame: every 30 minutes during hypothermia induction
Measure: Number; unit: participants
Arm/Group | Caffeinol
Number analyzed (Participants) | 30
participants | 0

ADVERSE EVENTS:
Time Frame: Adverse event data was collected over the duration of the study (2003-2009)
Arm/Group | Caffeinol
Serious Adverse Events (participants affected / at risk) | 9/30
Other Adverse Events (participants affected / at risk) | 17/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Caffeinol (N=30)
Death (Nervous system disorders) | 3 — Three patients died (SAE unrelated to study interventions): (1) symptomatic hemorrhage due to severity of stroke (1) malignant edema/ herniation (1) unrelated medical condition (withdrawal of care requested by family)
Neuroworsening (Nervous system disorders) | 4
Cholecysitits (Hepatobiliary disorders) | 1
Reduced respiratory drive (Respiratory, thoracic and mediastinal disorders) | 1
Parenchymal hemorrhage (Nervous system disorders) | 4 — 3 symptomatic 1 asymptomatic
Thrombotic thrombocytopenia (Blood and lymphatic system disorders) | 1 — Attributed to clopidrogrel and required treatment with plasmapheresis
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Caffeinol (N=30)
Sedation (Surgical and medical procedures) | 4 — Sedation noted: * (2)Demerol dose was reduced/held. Sedation resolved. * (2)Acidosis secondary to sedation. Treated/ resolved.
Elevated CK (Cardiac disorders) | 10 — Elevated Ck noted -asymptomatic/ resolved
Elevated Amylase (Gastrointestinal disorders) | 2 — Elevated amylase noted:Asymptomatic/resolved.
Device failure (Surgical and medical procedures) | 4 — Cooling machine failure (3) Icy catheter tubing leak (1)
Asymptomatic hemorrhagic transformation (Nervous system disorders) | 7 — Noted/ resolved
Elevated WBC (Blood and lymphatic system disorders) | 2 — No fever/ symptoms; resolved without treatment.
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 2 — (1)Treated with lasix and nebulizer treatment. Resolved. (1)Shortness of breath, oxygen saturation 87%, infiltrates on CXR. Treated with BiPAP & lasix
Infection (Infections and infestations) | 6 — * (2)UTI treated/ resolved. * GNR central line infection. Line removed/ antibiotic added. Resolved. * MRSA pneumonia treated. * Possible pneumonia treated with naficillin/ ceftin. * Pneumonia treated with antibiotics. Resolved.
Low Hgb/ Hct (Blood and lymphatic system disorders) | 2
Abnormal Labs (chem.) (Blood and lymphatic system disorders) | 3 — (1)Low K+ - replaced/ resolved (1)Elevated K+ - treated (1)Elevated Mg - asymptomatic/ resolved
Arrhythmia (Cardiac disorders) | 3 — (1) A. fib (1)A. fib with AV block
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes